CLINICAL TRIAL: NCT05353088
Title: Effects of Scapular Stabilization Versus Thoracic Spine Extension Exercises on Pain, Disability and Range Of Motion in Patients With Mechanical Neck Pain
Brief Title: Effects of Scapular Stabilization Versus Thoracic Spine Extension Exercises in Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0115 Anam
Record Dates: First submitted 2022-04-21; First posted 2022-04-29 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Neck Pain
Keywords: Disability Physical; muscle strength; range of motion
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapular stabilization exercises (Experimental): Group A performed scapular stabilization exercises for 4 weeks with 2 sets of 10 repetitions. These exercises comprised of four exercise programs (Scapular retraction; Scapular mobilization, Scapular dynamic stabilization I and Scapular dynamic stabilization II).
  Interventions: Other: scapular stabilization
- Thoracic extension exercises (Active Comparator): Group B performed thoracic extension exercises for 4 weeks with 2 sets of 10 repetitions. These exercises comprised of three exercise programs.
  Interventions: Other: Thoracic extension exercises

INTERVENTIONS:
Other: scapular stabilization — Scapular stabilization exercise aims to restore scapular position, orientations, motor control of muscles, and movement pattern, thereby attaining stability of scapula for better kinematics of shoulder.scapular stabilization exercises for 4 weeks with 2 sets of 10 repetitions. These exercises comprised of four exercise programs (Scapular retraction; Scapular mobilization, Scapular dynamic stabilization I and Scapular dynamic stabilization II)
  Arms: Scapular stabilization exercises
Other: Thoracic extension exercises — Thoracic extension involves concurrent posterior rotation (external torsion) and depression of the posterior ribs with elevation of the anterior ribs. Bending to the side is a combination of spinal segments side bending, ribs on the same come together while ribs on the opposite side separate.Group B performed thoracic extension exercises for 4 weeks with 2 sets of 10 repetitions. These exercises comprised of three exercise programs.
  Arms: Thoracic extension exercises

SUMMARY:
Mechanical neck pain is posteriorly occurring non-specific pain that originates from the superior nuchal line and extends to the first thoracic vertebrae. It is exacerbated by sustained neck postures, neck movements or cervical muscle palpation. The aim of study will be to compare the effects of scapular stabilization versus thoracic spine extension exercises on pain, disability and range of motion in patients with mechanical neck pain.

DETAILED DESCRIPTION:
A Randomized Clinical Trial will be conducted at Riphah Clinic Lahore, FMH Physiotherapy Clinic and Boston Physiotherapy Clinic Lahore through consecutive sampling technique on 30 patients which will be allocated using simple random sampling through sealed opaque enveloped into Group A and Group B. Group A will be treated with scapular stabilization exercises and Group B will be treated with thoracic extension exercises at the frequency of 2 sets with 10 repetitions and thrice a week. Outcome measures will be conducted through pain, disability and range of motion questionnaire after 6 weeks. Data will be analyzed during SPSS software version 21. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between 18 and 40 years of age with mechanical neck pain. (symptoms provoked by neck movement and/or palpation of musculature of the cervical region)
* Chronic mechanical neck pain for more than 3 months.

Exclusion Criteria:

* Cervical radiculopathy
* Traumatic neck injury
* History of cervical and thoracic spine surgery
* Neck pain associated with vertigo
* Osteoporosis
* Vertebral Fractures
* Tumors
* Pregnancy
* Diagnosed psychological disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | follow up at 6th week
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a unidimensional measure of pain intensity in adults, including those with chronic pain.
  The NPRS is a segmented numeric version in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain.
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
  The NPRS takes <1 minute to complete The NPRS is a valid and reliable scale to measure pain intensity;
  * High test-retest reliability has been (r = 0.96 and 0.95, respectively)
  * For construct validity, the NPRS was shown to be highly correlated: correlations range from 0.86 to 0.95.
Neck Disability index (NDI) | follow up at 6th week
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life. Every section is marked in each section only the one box that applies to you. We realise you may consider that two or more statements in any one section relate to you, but please just mark the box that most closely describes your problem. Intended population includes: Chronic neck or upper back pain and musculoskeletal neck pain.
  Scoring: For each section the total possible score is 5: if the first statement is marked the section score = 0, if the last statement is marked it = 5. If all ten sections are completed the score is calculated.
Range of Motion | follow up at 6th week
  A goniometer is an instrument that measures the available range of motion at a joint. To measure the range of motion physical therapists most commonly use a goniometer. It is necessary that a single notation system is used in goniometry. The neutral zero method (0 to 180- degree system) is the most widely used method. The same goniometer should always be used to reduce the chances of instrumental error.

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, MPhil, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Fatima memorial hospital - Physical therapy clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Korwisi B, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. Chronic pain as a symptom or a disease: the IASP Classification of Chronic Pain for the International Classification of Diseases (ICD-11). Pain. 2019 Jan;160(1):19-27. doi: 10.1097/j.pain.0000000000001384. PMID 30586067
- [Background] Masaracchio M, Kirker K, States R, Hanney WJ, Liu X, Kolber M. Thoracic spine manipulation for the management of mechanical neck pain: A systematic review and meta-analysis. PLoS One. 2019 Feb 13;14(2):e0211877. doi: 10.1371/journal.pone.0211877. eCollection 2019. PMID 30759118
- [Background] Gonzalez-Rueda V, Hidalgo-Garcia C, Rodriguez-Sanz J, Bueno-Gracia E, Perez-Bellmunt A, Rodriguez-Rubio PR, Lopez-de-Celis C. Does Upper Cervical Manual Therapy Provide Additional Benefit in Disability and Mobility over a Physiotherapy Primary Care Program for Chronic Cervicalgia? A Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Nov 11;17(22):8334. doi: 10.3390/ijerph17228334. PMID 33187167
- [Background] Mendes-Fernandes T, Puente-Gonzalez AS, Marquez-Vera MA, Vila-Cha C, Mendez-Sanchez R. Effects of Global Postural Reeducation versus Specific Therapeutic Neck Exercises on Pain, Disability, Postural Control, and Neuromuscular Efficiency in Women with Chronic Nonspecific Neck Pain: Study Protocol for a Randomized, Parallel, Clinical Trial. Int J Environ Res Public Health. 2021 Oct 12;18(20):10704. doi: 10.3390/ijerph182010704. PMID 34682453
- [Background] 5. Verma CV, Bhosale KS. Evaluation of neck pain and scapular stability in graduate dental students: A cross-sectional study. Indian Journal of Dental Sciences. 2021;13(4):260.
- [Background] Javdaneh N, Ambrozy T, Barati AH, Mozafaripour E, Rydzik L. Focus on the Scapular Region in the Rehabilitation of Chronic Neck Pain Is Effective in Improving the Symptoms: A Randomized Controlled Trial. J Clin Med. 2021 Aug 8;10(16):3495. doi: 10.3390/jcm10163495. PMID 34441791
- [Background] Yu L-J, Kim T-H. The Effect of Cervical Stabilization Exercises with Thoracic Spine Extension Exercises on Forward Head Posture. 2021.
- [Background] Seo YG, Park WH, Lee CS, Kang KC, Min KB, Lee SM, Yoo JC. Is Scapular Stabilization Exercise Effective for Managing Nonspecific Chronic Neck Pain?: A Systematic Review. Asian Spine J. 2020 Feb;14(1):122-129. doi: 10.31616/asj.2019.0055. Epub 2019 Nov 1. PMID 31668049
- [Background] Al-Bassiouny HA, Shendy S, El-Khozamy H. Effect of Upper Thoracic Mobilization on Chronic Mechanical Neck Pain. Med J Cairo Univ. 2019;87(3):1449-57.
- [Background] Yildiz TI, Turgut E, Duzgun I. Neck and Scapula-Focused Exercise Training on Patients With Nonspecific Neck Pain: A Randomized Controlled Trial. J Sport Rehabil. 2018 Sep 1;27(5):403-412. doi: 10.1123/jsr.2017-0024. Epub 2018 Jul 25. PMID 28605288